CLINICAL TRIAL: NCT00639704
Title: Evaluation of EM-IntraSPECT Reconstruction Algorithm by Comparison of Transmission Images Reconstructed From SPECT Projections Alone With MRI Studies
Brief Title: Improve Nuclear Medicine Heart Imaging, Compare MRI Results With Single Photon Emission Computed Tomography Imaging
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Andrzej Krol, PhD, State University of New York - Upstate Medical University
Other Study IDs: SUNYUMU 3257
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Cardiac
Keywords: MRI; SPECT; Cardiac function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the MRI results with the new SPECT image reconstruction method, this study will allow us to determine whether a new more accurate method of looking at the heart by nuclear study can be used in routine clinical use.

DETAILED DESCRIPTION:
Currently, up to one-third of all nuclear medicine studies are performed for cardiovascular disorders, and mostly are myocardial perfusion imaging (MPI) using SPECT acquisition. MPI aims at detection of acute myocardial ischemia and the scarred myocardium and it is increasingly used to plan myocardial revascularization and to assess the effectiveness of medical and surgical interventions. However, nonuniform gamma-ray attenuation in the thoracic region may severely impair the accuracy of SPECT cardiac imaging and frequently result in image artifacts. Therefore, attenuation corrected must be applied. We have derived an algorithm (called EM-IntraSPECT) that is able to reconstruct tomographic cross-sections of a patient from SPECT studies alone. The reconstructed cross-sections in turn, may be used for attenuation correction of cardiac SPECT images thus improving quality analysis based of these images. In this research we intend to continue evaluation of the new attenuation compensation algorithm and to assess the clinical usefulness of this method. These goals can be reached by comparing the patient's cross sectional anatomical data reconstructed by EM-IntraSPECT and obtained from MRI. It is proposed that 10 patients already undergoing nuclear cardiac imaging for clinical purpose, with 99mTc sestamibi or 99mTc radiolabeled red cells will be selected. These patients would be utilized to reconstruct transmission images and determination of internal anatomical structures in the thoracic region from SPECT projections alone. Further, direct and quantitative comparison of the patient's anatomy obtained by the MRI and the SPECT methods will be performed. The same algorithm would be used for reconstruction of attenuation compensated emission SPECT cardiac images. Finally, the accuracy and the clinical usefulness of this new, attenuation corrected cardiac SPECT image reconstruction would be quantitatively evaluated. All these procedures apply only to the image data and NOT the patient.

ELIGIBILITY:
Inclusion Criteria:

* subjects scheduled for cardiac SPECT
* subjects 18 years old or older

Exclusion Criteria:

* Females who are pregnant or think that they are pregnant will be excluded in this study.
* Subjects who have a pacemaker, internal defibrillator, prostheses, artificial heart valves, cardiac stents, surgical clips, or TENS (transcutaneous electric nerve stimulator)
* Subjects who are 300 lbs and over

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are being evaluated for cardiac function/perfusion
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 1996-01 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Krol, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States